CLINICAL TRIAL: NCT00558623
Title: Controlled Trial in Pregnancy of Dietary Supplements for Suppression of Bone Resorption and Mobilization of Lead Into Plasma
Brief Title: Dietary Calcium Supplementation to Reduce Blood Lead in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Collaborators: Mexican National Institute of Public Health (Other Government); Brigham and Women's Hospital (Other); University of California Santa Cruz (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P10345/9910CONT; NIEHS P42-ES05947 (Project 1)
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2007-11-15 (Estimated); Status verified 2007-11

CONDITIONS: Lead, Blood; Pregnancy; Bone Resorption
Keywords: lead, blood; pregnancy; calcium; randomized trial; dietary supplementation; bone resorption
MeSH Terms: conditions — Bone Resorption | interventions — Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: calcium carbonate

INTERVENTIONS:
Dietary Supplement: calcium carbonate — daily supplement of 1,200 milligrams calcium (two-600 mg tablets calcium carbonate at bedtime)
  Other Names: Lederle, Inc.

SUMMARY:
Lead accumulates in bone. During pregnancy, physiologic changes occur prompting bone resorption in order to provide calcium to the growing fetal skeleton also release the lead stored in bone into a pregnant woman's circulation. We have previously demonstrated that lead stores mobilized into the circulation of pregnant women pose a major threat to fetal development. This is particularly unfortunate since bone lead stores, once accumulated, persist for decades, thereby jeopardizing the pregnancies of women even if their current lead exposures have subsided. What then can be done for the many thousands of women who have had lead exposure while growing up and who want to have healthy children? To address this question, in 2000, this project embarked on a randomized intervention trial to test whether a bedtime nutritional supplement of 1,000 mg of calcium can significantly reduce fetal lead exposure and toxicity by suppressing bone resorption in the pregnant mother.

DETAILED DESCRIPTION:
Recent evidence indicates that there is a marked increase in the mobilization of lead from maternal bone stores into circulation during pregnancy and lactation. Furthermore, data from our group and others indicate that this phenomenon carries a significant risk of fetal toxicity in the form of growth (decreased birth weight, head circumference, birth length) and subsequent cognitive development. These findings pose a major public health problem, even among societies with declining lead exposure, given the persistence of pockets of high lead exposure (including some communities living in proximity to hazardous waste) as well as the long residence time of lead in bone (years to decades). One possible strategy for suppressing the mobilization of maternal bone lead stores during pregnancy is nutritional intervention. We are conducting a randomized, double-blinded, placebo-controlled trial of dietary supplements containing 1,200 milligrams of calcium as a means of suppressing bone resorption and the resulting mobilization of lead from bone into plasma during pregnancy, and into breast milk during the postpartum period. We are taking maternal measurements of pre-pregnancy and postpartum bone lead using our K-x-ray fluorescence technology; bone resorption (by assaying N-telopeptide of type I collagen in urine [urinary NTX]), whole blood lead, and plasma lead (using special collection techniques and measured by IDTIMS) during pre-pregnancy, the first, second, third trimesters and at one and four months postpartum; and breast milk lead levels at one and four months postpartum.

We are measuring maternal plasma and breast milk lead levels as these are the most direct sources of fetal and infant lead exposures, and recent research suggests that maternal venous blood lead levels do not adequately reflect either of these parameters. We are testing the hypothesis that supplements will significantly decrease urinary NTX, plasma lead, and breast milk lead levels. We are also exploring the relationship of plasma lead levels to birth anthropometry measures. This research, if successful, may provide a means of preventing secondary toxicity from accumulated lead burdens among women of reproductive age.

ELIGIBILITY:
Inclusion Criteria:

* being in the first trimester of pregnancy (no more than 14 weeks gestation); not presenting with a high-risk pregnancy; residing and plans to reside in the metropolitan Mexico City area for approximately 5 years; agreeing to participate and signing the informed consent form.

Exclusion Criteria:

* high-risk pregnancy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 670 (Actual)
Dates: Start 2001-01; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Blood Lead Concentration, Plasma Lead Concentration | 2nd, 3rd trimester pregnancy and 1,4,7,12 months postpartum

SECONDARY OUTCOMES:
Urinary Cross-linked N-telopeptides (marker of bone resorption) | 2nd, 3rd trimester of pregnancy and 1,4,7,12 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Howard Hu, MD, ScD, Principal Investigator — Harvard School of Public Health and University of Michigan; Mauricio Hernandez-Avila, MD, ScD, Principal Investigator — National Institute of Public Health and Ministry of Health, Mexico
Locations (1):
- Mauricio Hernandez-Avila, Cuernavaca, Morelos, Mexico

REFERENCES:
- [Derived] Perng W, Tamayo-Ortiz M, Tang L, Sanchez BN, Cantoral A, Meeker JD, Dolinoy DC, Roberts EF, Martinez-Mier EA, Lamadrid-Figueroa H, Song PXK, Ettinger AS, Wright R, Arora M, Schnaas L, Watkins DJ, Goodrich JM, Garcia RC, Solano-Gonzalez M, Bautista-Arredondo LF, Mercado-Garcia A, Hu H, Hernandez-Avila M, Tellez-Rojo MM, Peterson KE. Early Life Exposure in Mexico to ENvironmental Toxicants (ELEMENT) Project. BMJ Open. 2019 Aug 26;9(8):e030427. doi: 10.1136/bmjopen-2019-030427. PMID 31455712
- [Derived] Ettinger AS, Lamadrid-Figueroa H, Mercado-Garcia A, Kordas K, Wood RJ, Peterson KE, Hu H, Hernandez-Avila M, Tellez-Rojo MM. Effect of calcium supplementation on bone resorption in pregnancy and the early postpartum: a randomized controlled trial in Mexican women. Nutr J. 2014 Dec 16;13(1):116. doi: 10.1186/1475-2891-13-116. PMID 25511814